CLINICAL TRIAL: NCT03649659
Title: Phase III RCT of the Effectiveness of Silver Diamine Fluoride in Arresting Cavitated Caries Lesions
Brief Title: Effectiveness of Silver Diamine Fluoride (SDF) in Arresting Cavitated Caries Lesions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial stopped early due to meeting interim analysis early stopping rules. Active participants at the time of the interim analyses results did complete their remaining study visits. No new participants were enrolled.
Sponsor: University of Michigan (Other)
Collaborators: NYU Langone Health (Other); University of Iowa (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Margherita Fontana, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00147622; U01DE027372 (NIH)
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Cavities of Teeth
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (SDF) (Experimental): SDF will be applied to the affected teeth twice during the study. Once at screening/baseline and again at the 6-month visit.
  Interventions: Drug: Silver Diamine Fluoride
- Placebo (Placebo Comparator): The placebo will be applied to the affected teeth twice during the study. Once at screening/baseline and again at the 6-month visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silver Diamine Fluoride — SDF will be applied twice during the study
  Other Names: Diammine Silver Fluoride
  Arms: Silver Diamine Fluoride (SDF)
Drug: Placebo — This is being compared to the SDF and will also be applied twice
  Arms: Placebo

SUMMARY:
This trial is a Phase III, multisite, randomized, placebo-controlled trial, with two parallel groups. The groups are SDF or placebo and they are applied every 6 months. The primary hypothesis of the trial is that SDF is better than placebo for stopping cavities with dentin exposed in baby teeth when assessed at 6 months after initial application.

DETAILED DESCRIPTION:
This trial is a phase III, multicenter, randomized, placebo-controlled superiority trial, with two parallel groups (placebo vs. SDF applied to cavitated lesions) involving a total of 1144 children with the primary outcome assessed at 6 months after initial treatment.

One thousand one hundred forty four children, 12-71 months of age, from early childhood education programs, such as Head Start centers, Early Head Start centers, and equivalent city/state subsidized preschool programs, or children attending dental clinics associated with the clinical trial sites, will be randomized, in two cohorts. Trial visits will occur at baseline, 3 months, 6 months, and 8 months. SDF/placebo will be applied at baseline and 6 months. Parents/legal guardians will be called 24 to 48 hours after the SDF/placebo application to assess adverse events and unanticipated problems and in-person visits for safety exams will be available for all child participants approximately 24 to 48 hours after SDF/placebo application. This visit could happen before or after the 24- to 48-hour call with the parent or legal guardian, but every attempt will be made so that the call occurs prior to the 24- to 48-hour visit. Additionally, intermediate contacts at 1.5 months, 4.5 months, and 7 months will occur to determine if the child needs an additional visit to assess pain, lesion progression, etc. and to maintain contact with the participant.

Randomization to SDF application (treatment) or placebo (control) will be at the participant-level; all teeth within a participant that meet the inclusion criteria will receive the same trial product. Both treatment and control will be dispensed from identical unit-dose ampules coded and labeled to ensure masking of all trial personnel. The number of ampules required to treat all carious lesions in the participant's mouth will be recorded. No caries removal will be performed. Teeth will be cleaned with a toothbrush and will be dried with cotton/gauze, and the solution will be painted on the dentin of each targeted cavitated lesion using a standardized applicator. Following application, the tooth will be blotted dry with gauze.

At each clinical visit International Caries Detection and Assessment System (ICDAS) examinations, including cavitated lesion hardness assessments, soft tissue assessments and questionnaires on dental discomfort, family impact and treatment satisfaction and acceptability will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Child:

  * Male or female, between 12-71 months of age at baseline, up to the day the child turns 6 years old.
  * Must allow examination of the oral cavity and application of treatment by the examiners at baseline.
  * Must have S-ECC [defined as: In children younger than age 3, any sign (non-cavitated or cavitated lesion) of caries in any tooth surface (i.e., most common for this age group will be on erupted smooth surfaces). From ages 3 through 5, ≥1 dmfs in maxillary anterior teeth; or a dmfs score of ≥4 (age 3), ≥5 (age 4), or ≥6 (age 5) constitutes S-ECC. Note: The "d" component of the dmfs index is defined as including cavitated and non-cavitated lesions, thus ICDAS>1].
  * Have at least one SDF-target tooth with

    * Soft cavitated caries lesions extending into dentin [ICDAS 5 or 6];
    * Cavitated lesion(s) that allow for direct hardness assessment and application of SDF (microbrush applicator must fit the cavity and be able to access all exposed dentin).
* Parent/Legal Guardian:

  * Provide written informed consent for the child and her/himself prior to participation.
  * Must be at least 18 years old, or an emancipated minor who provides documentation of emancipation.
  * Must be willing and able to participate in trial activities.

Exclusion Criteria:

* Child:

  * Hereditary generalized developmental dental defects such as Amelogenesis Imperfecta and Dentinogenesis Imperfecta.
  * Known allergy/sensitivity to silver or other heavy metal ions.
  * Presence of any gingival or peri-oral ulceration, abscess or stomatitis.
  * Participating in the foster care system at trial initiation.
  * Toothache pain at baseline (based on Dental Discomfort Questionnaire score of 1 or higher).

    * Note: If toothache pain occurs after baseline, the child remains eligible to continue in the trial as long as he/she has at least one trial tooth that meets tooth inclusion/exclusion criteria.
  * Demonstrated inability to comply with trial protocol requirements (determination is at the Clinical Site Investigator's discretion).
  * Rickets.
  * Osteopenia or osteoporosis (e.g., Osteogenesis Imperfecta, Ehlers-Danlos Syndrome, Marfan Syndrome, etc.).
  * Chronic diseases such as chronic kidney disease, leukemia, lymphoma, rheumatic disorders, etc.
  * Metabolic bone disease (e.g., Galactosemia, Glycogen Storage Disease Type 1, etc.).
  * Chronic glucocorticoid, anticonvulsants, chemotherapy, bisphosphonate administration.
  * Hypothyroidism, hyperparathyroidism, impaired glucose tolerance, hypocalcemia or hypophosphatemia.
* Tooth:

  * Pain due to caries (based on DDQ score of 1 or higher).

    * Note: If toothache pain occurs after baseline, the tooth is removed from the study.
  * Pulpal exposure, or signs of pulpal infection (abscess, fistula, swelling).
  * Mobility not associated with expected exfoliation patterns.
* Parent/Legal Guardian:

  * Demonstrated inability to comply with trial protocol requirements (determination is at the Clinical Site Investigator's discretion).
  * Inability to read and comprehend the consent document or trial questionnaires in the translated languages available.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 830 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margherita Fontana, DDS, PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Iowa College of Dentistry, Iowa City, Iowa
  - University of Michigan School of Dentistry, Ann Arbor, Michigan
  - New York University College of Dentistry, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
Started | 414 | 416
Completed | 278 | 265
Not Completed | 136 | 151

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo | Total
Number analyzed (Participants) | 414 | 416 | 830
Age, Customized [Count of Participants; unit: Participants]
  Child Age 1 Years | 15 | 19 | 34
  Child Age 2 Years | 56 | 56 | 112
  Child Age 3 Years | 124 | 107 | 231
  Child Age 4 Years | 155 | 170 | 325
  Child Age 5 Years | 64 | 64 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 200 | 428
  Male | 186 | 216 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 182 | 183 | 365
  Not Hispanic or Latino | 228 | 219 | 447
  Unknown or Not Reported | 4 | 14 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 26 | 24 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 86 | 171
  White | 138 | 132 | 270
  More than one race | 24 | 37 | 61
  Unknown or Not Reported | 138 | 134 | 272
Region of Enrollment [Number; unit: participants]
  United States | 414 | 416 | 830

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Arrested Trial Lesions Per Child in Each Treatment Arm After One Treatment With SDF or Placebo
Description: Arrested trial lesions will be assessed by determining if the lesion is hard or soft by pressing on the lesion using a standard probe as assessed by calibrated examiners.
Time Frame: 6 months
Measure: Mean (99.9% Confidence Interval); unit: percentage of lesions arrested
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
Number analyzed (Participants) | 414 | 416
percentage of lesions arrested | 54 [43.1 to 64.4] | 22.5 [15.3 to 31.8]
Statistical Analysis 1: Comparison: Silver Diamine Fluoride (SDF) vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Multiple imputation (25) of missing data, FCS methods. Group comparisons using GEE logistic model, exchangeable correlation, study site as covariate; Odds Ratio (OR) = 4.06, 99.9% CI 2-sided [2.54 to 6.48]

2. Secondary Outcome: The Proportion of Arrested Trial Lesions Per Child in Each Treatment Arm After Two Treatments With SDF or Placebo
Description: Arrested trial lesions will be assessed by determining if the lesion is hard or soft after two SDF applications by pressing on the lesion using a standard probe as assessed by calibrated examiners.
Time Frame: 8 months
Measure: Mean (99.9% Confidence Interval); unit: percentage of lesions arrested
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
Number analyzed (Participants) | 414 | 416
percentage of lesions arrested | 50.2 [39.5 to 60.9] | 17.4 [11.4 to 25.7]
Statistical Analysis 1: Comparison: Silver Diamine Fluoride (SDF) vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic — Multiple imputation (25) of missing data, FCS methods. Group comparisons using GEE logistic model, exchangeable correlation, study site as covariate; Odds Ratio (OR) = 4.78, 99.9% CI 2-sided [2.84 to 8.05]

3. Secondary Outcome: Proportion of Arrested Trial Lesions Per Child in Each Treatment Arm After One Treatment With SDF or Placebo
Description: Proportion of arrested trial lesions will be assessed by determining if the lesion is hard or soft by pressing on the lesion using a standard probe as assessed by calibrated examiners. The effect of a single application will be assessed at 3-month follow-up post initial treatment.
Time Frame: 3 months
Measure: Mean (99.9% Confidence Interval); unit: percentage of lesion arrest
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
Number analyzed (Participants) | 414 | 416
percentage of lesion arrest | 57.5 [46.5 to 67.8] | 18.8 [12.4 to 27.5]
Statistical Analysis 1: Comparison: Silver Diamine Fluoride (SDF) vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.84, 99.9% CI 2-sided [3.59 to 9.51]

4. Secondary Outcome: Proportion of Trial Lesions With Pain Prior to or at the 8-month Visit
Description: The presence of pain associated with a trial lesion was screened at baseline a score of 1 or higher using the Dental Discomfort Questionnaire (DDQ). The DDQ is a validated tool assessing pain in children 5 and younger, as reported by parents/legal guardians, based on observation of toothache pain-related behaviors by the child. It consists of two parts: a question of the occurrence of toothache and when (if no pain DDQ score of 0,best), and 8 validated questions about behaviors associated with toothache or discomfort due to caries on a three-point scale: 0 'never', 1 'sometimes', and 2 'often'. Total score is the sum of the 8 questions in part two, ranging from 0 (no pain) to 16 (worst score). A DDQ score of 1 or higher may not be caused by pain in a trial tooth, so children with a DDQ score of 1 or higher were examined during a clinical visit to determine if the trial teeth had pain. Pain associated with a trial tooth at any time after baseline treatment counted as trial lesion pain.
Time Frame: Baseline, 24-48 hour call, 1.5 month, 3 month, 4.5 month, 6 month, 24-48 hours after 6 month, 7 month, 8 month
Measure: Mean (99.9% Confidence Interval); unit: percentage of trial lesions with pain
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
Number analyzed (Participants) | 414 | 416
percentage of trial lesions with pain | 2.7 [0.8 to 8.9] | 2.8 [0.8 to 9.6]
Statistical Analysis 1: Comparison: Silver Diamine Fluoride (SDF) vs Placebo; Test type: Superiority; p = 0.8942, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.95, 99.9% CI 2-sided [0.25 to 3.54]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Silver Diamine Fluoride (SDF) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/414 | 0/416
Serious Adverse Events (participants affected / at risk) | 3/414 | 1/416
Other Adverse Events (participants affected / at risk) | 103/414 | 89/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silver Diamine Fluoride (SDF) (N=414) | Placebo (N=416)
Hospitalization for Dental Abscess (Gastrointestinal disorders) | 1 | 0 — Hospitalization due to infection and pain with dental abscess resulting in tooth extraction
Hospitalization for Appendix Removal (Surgical and medical procedures) | 1 | 0 — Inpatient stay for surgical removal of appendix due to diagnosis of appendicitis.
Hospitalization for Febrile Seizure (General disorders) | 1 | 0 — Cough and fever and subsquent febrile seizure resulting in hospital admission for two nights to stabilize.
Hospitalization due to Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Abnormal breathing resulting in hospital admission for two nights to diagnose and stabilize. Diagnosis of chronic asthma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silver Diamine Fluoride (SDF) (N=414) | Placebo (N=416)
Abscess (Gastrointestinal disorders) | 35 | 34
Allergic Reaction (Immune system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dental Trauma (Injury, poisoning and procedural complications) | 2 | 2
Dental Treatment (Surgical and medical procedures) | 22 | 18
Diarrhea (Gastrointestinal disorders) | 3 | 0
Ear Infection (Infections and infestations) | 3 | 5
Extraoral Staining (Injury, poisoning and procedural complications) | 5 | 0
Fever (General disorders) | 9 | 16
Gastrointestinal Pain (Gastrointestinal disorders) | 4 | 4
Intraoral Staining (Injury, poisoning and procedural complications) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oral Erythema (Gastrointestinal disorders) | 2 | 1
Oral Pain (Gastrointestinal disorders) | 1 | 3
Oral Ulceration (Gastrointestinal disorders) | 1 | 2
Other (General disorders) | 15 | 6 — COVID-19, heatstroke, dog bite, halitosis, muscle pain, congestion, cheek swelling, seasonal allergies, self-reported flu, stye, helicobacter pylori
Other Surgical Procedure (Surgical and medical procedures) | 1 | 2 — Tonsillectomies, ear tube surgeries, staples, stitches
Pulpal Exposure (Gastrointestinal disorders) | 6 | 8
Respiratory Infection (Infections and infestations) | 7 | 8
Skin and Tissue Disorders (Skin and subcutaneous tissue disorders) | 6 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 33 | 26
Vomiting (Gastrointestinal disorders) | 5 | 8

LIMITATIONS AND CAVEATS:
The trial was stopped early due to efficacy after the interim analysis. All subjects enrolled when the early termination was decided were allowed to finish the trial and their data were included in the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03649659/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03649659/SAP_003.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT03649659/ICF_002.pdf